CLINICAL TRIAL: NCT00362297
Title: A Randomized, Cross-Over Study to Evaluate the Suppressive Effect of High-Dose Acyclovir Versus Once Daily Valacyclovir on Herpes Simplex Virus Type 2 Genital Shedding in Herpes Simplex Virus-2 Seropositive Adults
Brief Title: Randomized Trial to Evaluate Suppressive Effect of High-Dose Acyclovir Versus Once-Daily Valacyclovir on Persons With HSV-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Christine Johnston, Acting Assistant Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 30520-D - Phase 1
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Genital Herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — Acyclovir; Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dose (Active Comparator)
  Interventions: Drug: valacyclovir
- High-dose (Experimental)
  Interventions: Drug: acyclovir

INTERVENTIONS:
Drug: acyclovir — 800 mg orally three times daily for 7 weeks
  Arms: High-dose
Drug: valacyclovir — 500 mg orally once daily for 7 weeks
  Other Names: Valtrex
  Arms: Standard dose

SUMMARY:
The purpose of the research study is to evaluate the effectiveness of high-dose acyclovir compared to valacyclovir for reduction of asymptomatic genital shedding in persons with genital herpes.

The study will enroll men and women who are 18 years or older, test positive to HSV-2 (by blood test) and have had a first outbreak of HSV-2 within the past 6 months or have had at least 4 genital herpes outbreaks in the past year. Participants must be HIV negative and willing to stop taking suppressive therapy for HSV for the one week wash out period. (Females only: You must not be pregnant or breast-feeding). Both men and women will be asked to use an effective form of birth control.

Involvement in the study will last 15-weeks and you will be asked to visit the clinic every 2-weeks. At each visit, you will be given medication to take daily (either valacyclovir or acyclovir; you will receive both medications at some point during this study). There will be a total of 9 study visits and each visit will last approximately 30 minutes. We will ask that you complete a daily symptom diary and collected daily home swabs 4-times a day, everyday during the study. Each daily home swab will take less than 3 minutes to perform.

DETAILED DESCRIPTION:
Screening Assessment

Patients will be assessed for their eligibility to enter the study at a screening visit. After signing informed consent they will undergo a medical history and the following information will be recorded in the Case Report Form (CRF):

* Demographic Data: Date of birth, sex, marital status, education and race
* Previous antiviral medication taken
* History of sexually transmitted infections and sexual history.

Start of Study Visit (Day 0) and Day 14, 28, 42, 56, 70, 84, 98 and 105 Follow-Up Visits.

Eligible patients will return to clinic to be given study drug and a patient diary card on which to record concomitant medications, signs and symptoms, and adverse experiences. The investigator will instruct the patient on daily home viral sample collection, taking the study drug, and completing the diary card. The patient will be instructed to return to clinic in 2 weeks, +/- 2 days. Medication compliance will be assessed at each visit using pill counts.

Crossover Study Visit Prior To Washout Period (Day 49-55)

Participants will not be given study drug or placebo during the 7-day washout period.

Daily Home Viral Sample Collection

Participants will collect swabs from the genital mucosa four times per day and store the samples in PCR media with preprinted labels. Women will swab the cervicovaginal, vulvar and perianal areas, and men will swab the penile and perianal. Every two weeks, they will return the samples to the Virology Research Clinic when they present for additional study drug and assessment.

Final Study Visit (Day 105)

At the final study visit at Day 105 or for premature discontinuation, the investigator will perform the activities at the regular study visits, with the exception of the dispensation of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older;
2. HSV-2 seropositive by Western Blot;
3. not receiving any drugs with known anti-HSV-2 activity for study duration;
4. history of primary genital herpes infection within past 6 months OR history of 4 or more HSV recurrences per year during the past year OR 4 or more recurrences per year prior to initiation of suppressive antiviral therapy;
5. able to comply with the study protocol;
6. women of child bearing potential who are sexually active with men must be using a medically accepted method of contraception as judged by the investigator;
7. women of child-bearing potential must have a negative pregnancy test (urine) at screening visit;
8. in general good health, without other serious medical conditions and specifically with normal renal and hepatic function, as determined by the patient's medical history;
9. planning to remain resident in the area of the study center for the duration of the study participation;
10. HIV seronegative.

Exclusion Criteria:

1. hypersensitivity to acyclovir or valacyclovir;
2. pregnant women;
3. HIV positive or other immunosuppressed state, including chronic steroid use. Intermittent nasal or topical steroids are acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Johnston, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States

REFERENCES:
- [Derived] Johnston C, Saracino M, Kuntz S, Magaret A, Selke S, Huang ML, Schiffer JT, Koelle DM, Corey L, Wald A. Standard-dose and high-dose daily antiviral therapy for short episodes of genital HSV-2 reactivation: three randomised, open-label, cross-over trials. Lancet. 2012 Feb 18;379(9816):641-7. doi: 10.1016/S0140-6736(11)61750-9. Epub 2012 Jan 4. PMID 22225814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: November 2006-August 2008 Site: University of Washington Virology Research Clinic, Seattle, WA
Period: Treatment 1 (Initial Drug Assignment)
Arm/Group | Standard Dose First, Then High Dose | High Dose First, Then Standard Dose
Started | 16 | 15
Completed | 16 | 11
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 4
Period: Treatment 2
Arm/Group | Standard Dose First, Then High Dose | High Dose First, Then Standard Dose
Started | 16 | 11
Completed | 16 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose | High-dose | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (13.2) | 39.1 (12.2) | 40.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 13 | 10 | 23
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Frequency of HSV-2 Total Shedding From the Genital Tract as Measured by PCR, Calculated Using a Per-day Shedding Rate in Participants Treated With High-dose Acyclovir as Compared to Once-daily Valacyclovir.
Description: Participants were treated with both interventions in a cross-over study design. Shedding rates on each drug arm per participant were compared by Poisson regression. Shedding rates were calculated by dividing the number of positive swabs by the total number of swabs for each intervention group.
Time Frame: 15 weeks
Population: Participants who did not collect at least one swab on each arm of the cross-over were excluded from analysis.
Measure: Number; unit: percentage of swabs with HSV detected
Units Other Than Participants: Swabs
Arm/Group | Standard Dose Valacyclovir | High Dose Acyclovir
Number analyzed (Participants) | 27 | 27
Number analyzed (Swabs) | 4663 | 4709
percentage of swabs with HSV detected | 4 | 4
Statistical Analysis 1: Comparison: Standard Dose Valacyclovir; Comparison of genital HSV shedding rate on high dose acyclovir to standard dose valacyclovir. Powered with 80% chance of detecting 50% reduction in genital shedding rate on high dose acyclovir compared to standard dose valacyclovir; Test type: Superiority or Other; p = 0.052, Regression, Poisson; Adjusted for period effects; Incident Risk Ratio = 0.79, 95% CI [0.63 to 1.00]

ADVERSE EVENTS:
Arm/Group | Standard Dose | High-dose
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/31
Other Adverse Events (participants affected / at risk) | 0/27 | 0/31

LIMITATIONS AND CAVEATS:
The trial was performed at a single site, and enrolled mostly white, healthy, sexually active adults with high rates of genital HSV-2 recurrence. The results may not be generalizable to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No